CLINICAL TRIAL: NCT02170272
Title: Development and Pilot Testing of a Home-Based Program for Head and Neck Cancer Survivors With Lymphedema
Brief Title: Home-Based Lymphedema Care Program (HBLCP) in Improving Lymphedema Self-Care in Head and Neck Cancer Survivors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to obtain funding
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Vanderbilt Office of Clinical and Translational Scientist Development (Unknown)
Responsible Party: Principal Investigator, Jie Deng, Principal Investigator, Vanderbilt-Ingram Cancer Center, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VICC HN 1431; NCI-2014-00867 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA068485 (NIH)
Record Dates: First submitted 2014-06-13; First posted 2014-06-23 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Head and Neck Cancer; Lymphedema
MeSH Terms: conditions — Head and Neck Neoplasms; Lymphedema | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Home-based Lymphedema Care Program (Experimental): Home-based Lymphedema Care Program (HBLCP): Participants will undergo one training session with a lymphedema therapist, and then receive a self-care video and educational manual to review at home. After completion of training session, follow-up measures occur at 1, 2, and 3 months.
  Interventions: Behavioral: Home-based Lymphedema Care Program

INTERVENTIONS:
Behavioral: Home-based Lymphedema Care Program — Undergo HBLCP
  Other Names: intervention, educational

SUMMARY:
This pilot clinical trial studies a home-based lymphedema care program in improving lymphedema self-care in head and neck cancer survivors. A home-based lymphedema care program may help head and neck cancer survivors manage their lymphedema and improve their well-being and quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop a home-based lymphedema care program (HBLCP) focusing on self-care of head and neck lymphedema in head and neck cancer (HNC) patients who have received lymphedema therapy. (Stage 1) II. To assess feasibility of the HBLCP for HNC patients with lymphedema to: 1) obtain recruitment estimates and determine barriers to recruitment; 2) evaluate implementation fidelity (i.e., competence and compliance) and barriers to implementation fidelity; 3) assess safety; and 4) evaluate satisfaction. (Stage 2) III. To obtain preliminary efficacy data of the HBLCP via the following indicators: 1) head and neck lymphedema; 2) symptom burden; and 3) functional status. (Stage 2)

OUTLINE:

INTERVENTION DEVELOPMENT: A team of experts complete the development of a patient self-care video, an educational manual, a therapist training video, and a protocol. Lymphedema therapists test the therapist training video and protocol. Patients then undergo a training session with the study therapy and test the patient video and educational manual.

PILOT HBLCP TESTING: Participants undergo one training session with a lymphedema therapist. Participants also receive a self-care video and educational manual to review at home.

After completion of training session, participants are followed up at 1, 2, and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* STAGE 1:
* EXPERT PANEL:
* A convenience sample of 10-15 experts (at least three lymphedema therapists and a varying number of HNC medical, radiation, and surgical oncologists, HNC nurse practitioners, speech and language pathologists, and nursing and informatics scientists) will be recruited to inform development of videos, protocol, and educational manual
* Knowledgeable in either HNC or lymphedema management or informatics
* LYMPHEDEMA THERAPISTS:
* Subsequent to the development of the materials, five additional therapists will be recruited to conduct an unbiased test of the therapists' training video and protocol
* Certified lymphedema therapists
* Knowledgeable in head and neck lymphedema management
* PATIENT PARTICIPANTS:
* A convenience sample of 10 HNC survivors will be recruited to undergo a training session with the study therapist and test the patient video and educational manual
* Post HNC primary treatment
* No evidence of cancer (NED)
* Completion of lymphedema therapy for lymphedema of the head and neck
* Ability to understand English in order to complete questionnaires
* Able to complete the onsite training and home self-care activities for lymphedema management
* Able to provide informed consent
* STAGE 2 PATIENT PARTICIPANTS:
* Using the same inclusion criteria as Stage 1 a convenience sample of 30 different HNC survivors will be recruited

Exclusion Criteria:

* Patients with medical conditions (e.g., acute infection, congestive heart failure, renal failure, cardiac or pulmonary edema, sensitive carotid sinus, severe carotid blockage, and uncontrolled hypertension) that would prohibit the safe implementation of home-based self-care of lymphedema will be excluded

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change in severity rate of head and neck lymphedema | Baseline to up to 3 months
  Compared to baseline, head and neck cancer survivors with lymphedema who participates in the HBLCP will have improved outcome (e.g., decreased lymphedema severity) through measures of CTCAE, External HNLE-Fibrosis Grading Criteria, and Foldi's Scale at the study follow-ups

SECONDARY OUTCOMES:
Change in rating of severity symptom burden | Baseline to up to 3 months
  Compared to baseline, head and neck cancer survivors with lymphedema who participates in the HBLCP will have improved outcome (e.g., decreased symptom burden) through measures of VHNSS and LSIDS-H&N at the study follow-ups
Change in rating of jaw, neck, and shoulder range of motion | Baseline to up to 3 months
  Compared to baseline, head and neck cancer survivors with lymphedema who participates in the HBLCP will have improved functional outcome measures in jaw, neck, and shoulder range of motion at the study follow-ups

OTHER OUTCOMES:
Assessment of feasibility of the HBLCP for head and neck cancer survivors with lymphedema | Baseline to up to 3 months
  The major measures include to: 1) determine barriers to recruitment; and 2) evaluate implementation fidelity (i.e., competence and compliance) and barriers to implementation fidelity through feasibility questionnaires.
Recruitment estimates through number of patients recruited | Up to 3 months
  Recruitment Log will be used to document recruitment information

CONTACTS AND LOCATIONS:
Overall Officials: Jie Deng, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/